CLINICAL TRIAL: NCT06130709
Title: IRAF-ABLATION Study: a Multicenter International Retrospective Cohort of Patients With BTK Inhibitors-related AF Treated by Catheter Ablation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: IRAF-Ablation
Record Dates: First submitted 2023-11-06; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: BTKi-induced Atrial Fibrillation; Hematologic Malignancy; Atrial Fibrillation Catheter Ablation
Keywords: atrial fibrillation; Bruton tyrosine kinase inhibitors; catheter ablation,; atrial fibrillation recurrence
MeSH Terms: conditions — Hematologic Neoplasms; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Atrial fibrillation catheter ablation in a population of BTKi-induced atrial fibrillation — Atrial fibrillation catheter ablation in a population of BTKi-induced atrial fibrillation

SUMMARY:
Targeted anticancer drugs have completely changed the prognosis of malignancies during the past decades. Patients suffering from malignancies live longer and this allows adverse events of anticancer drugs to emerge, notably cardiovascular adverse events. It is particularly important because of the great morbimortality of major cardiovascular events like myocardial infarction or stroke and because of their frequency in cancer populations. Indeed, cardiovascular death is the second cause of deaths after malignancy itself in this population. Atrial fibrillation (AF) is a non rare cardiovascular adverse events associated with a shorter overall survival in some malignancies localization. The emblematic anticancer drugs promoting AF is ibrutinib belonging to the Bruton tyrosine kinase inhibitors (BTKi), which are indicated in hematological malignancies. Incidence of AF with ibrutinib is estimated to 4.92/100 person-years; 95% CI: 2.91-4.81 but is underestimated because of the absence of systematic electrocardiogram recording. The management of AF rests on anticoagulation if indicated by the CHA2DS2-VASc score, and on the choice between a rate or rhythm control strategy. Rate control is the privileged strategy because of the risk of drugs interactions of the anti-arrhythmic drugs in a context of anticancer drugs co-prescriptions. But in case of symptoms with normal heart rate, life expectancy counted in years and preserved condition, catheter ablation has to be discussed. Whereas this interventional procedure has been greatly studied in the general population, no study exists in patients with hematological malignancies. The investigators aim to describe baseline characteristics of a population of BTKi-induced AF undergone AF catheter ablation.

DETAILED DESCRIPTION:
Targeted anticancer drugs have completely changed the prognosis of malignancies during the past decades. Patients suffering from malignancies live longer and this allows adverse events of anticancer drugs to emerge, notably cardiovascular adverse events. It is particularly important because of the great morbimortality of major cardiovascular events like myocardial infarction or stroke and because of their frequency in cancer populations. Indeed, cardiovascular death is the second cause of deaths after malignancy itself in this population. Atrial fibrillation (AF) is a non rare cardiovascular adverse events associated with a shorter overall survival in some malignancies localization. The emblematic anticancer drugs promoting AF is ibrutinib belonging to the Bruton tyrosine kinase inhibitors (BTKi), which are indicated in hematological malignancies. Incidence of AF with ibrutinib is estimated to 4.92/100 person-years; 95% CI: 2.91-4.81 but is underestimated because of the absence of systematic electrocardiogram recording. The management of AF rests on anticoagulation if indicated by the CHA2DS2-VASc score, and on the choice between a rate or rhythm control strategy. Rate control is the privileged strategy because of the risk of drugs interactions of the anti-arrhythmic drugs in a context of anticancer drugs co-prescriptions. But in case of symptoms with normal heart rate, life expectancy counted in years and preserved condition, catheter ablation has to be discussed. Whereas this interventional procedure has been greatly studied in the general population, no study exists in patients with hematological malignancies. The investigators aim to describe baseline characteristics of a population of BTKi-induced AF undergone AF catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* every adult patient treated by BTKi for a hematological malignancy
* with a new onset recurrence of AF occurring after BTKi initiation and treated by catheter ablation
* with an available 12 months follow up after catheter ablation

Exclusion Criteria:

* Patients younger than 18 years old
* Severe mitral regurgitation/stenosis or rhumatismal heart disease whatever the grade
* Permanent AF
* Patient who had AF rhythm during the first administration of BTKi

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population treated with iBTK for hematologic malignancy and who developped BTKi-induced atrial fibrillation treated by cathter ablation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Description of the one-year AF recurrence rate after catheter ablation in a population of BTKi induced AF | 1 year follow-up from the catheter ablation date
  AF recurrence is defined as atrial fibrillation or atrial tachycardia or atrial flutter, on a single 12-lead ECG or lasting more than 30 seconds on Holter monitoring in the period between the end of the 3-month blanking period and 12-month follow-up.

SECONDARY OUTCOMES:
Description of the baseline characteristic of the population of BTKi induced AF with AF catheter ablation carried out | At inclusion (= the time of ablation date)
Description of atrial electrophysiological properties during AF catheter ablation in a population of BTKi induced AF | At inclusion (= the time of ablation date)
Description of AF catheter ablation complications at 3 months follow-up in a population of BTKi induced AF (MACE, sepsis, bleeding, hospitalization prolongation, hospitalization readmission, mortality) | 3 months follow-up from the ablation date
Identification of baseline parameters and electrophysiologic parameters associated with AF recurrence at 12 months follow-up | 1 year follow-up from the catheter ablation date

CONTACTS AND LOCATIONS:
Overall Officials: Joachim ALEXANDRE, MD, PhD, Principal Investigator — Caen Normandy University Hospital, France
Locations (1):
- Caen University Hospital, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandre J, Salem JE, Moslehi J, Sassier M, Ropert C, Cautela J, Thuny F, Ederhy S, Cohen A, Damaj G, Vilque JP, Plane AF, Legallois D, Champ-Rigot L, Milliez P, Funck-Brentano C, Dolladille C. Identification of anticancer drugs associated with atrial fibrillation: analysis of the WHO pharmacovigilance database. Eur Heart J Cardiovasc Pharmacother. 2021 Jul 23;7(4):312-320. doi: 10.1093/ehjcvp/pvaa037. PMID 32353110
- [Background] Lyon AR, Lopez-Fernandez T, Couch LS, Asteggiano R, Aznar MC, Bergler-Klein J, Boriani G, Cardinale D, Cordoba R, Cosyns B, Cutter DJ, de Azambuja E, de Boer RA, Dent SF, Farmakis D, Gevaert SA, Gorog DA, Herrmann J, Lenihan D, Moslehi J, Moura B, Salinger SS, Stephens R, Suter TM, Szmit S, Tamargo J, Thavendiranathan P, Tocchetti CG, van der Meer P, van der Pal HJH; ESC Scientific Document Group. 2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS). Eur Heart J. 2022 Nov 1;43(41):4229-4361. doi: 10.1093/eurheartj/ehac244. No abstract available. PMID 36017568
- [Result] Agarwal S, Munir MB, Krishan S, Yang EH, Barac A, Asad ZUA. Outcomes and readmissions in patients with cancer undergoing catheter ablation for atrial fibrillation. Europace. 2023 Aug 2;25(9):euad263. doi: 10.1093/europace/euad263. No abstract available. PMID 37655932